CLINICAL TRIAL: NCT00333216
Title: Efficacy and Safety of Posterior Juxtascleral Administrations of Anecortave Acetate for Depot Suspension (15 mg or 30 mg) Versus Sham Administration in Singaporean Patients at Risk for Progressing to Exudative Age-Related Macular Degeneration (AMD)
Brief Title: Anecortave Acetate Risk-Reduction Trial (AART)
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Lack of efficacy
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: C-04-30
Record Dates: First submitted 2006-05-31; First posted 2006-06-02 (Estimated); Last update posted 2012-11-28 (Estimated); Status verified 2011-12

CONDITIONS: AMD
MeSH Terms: interventions — anecortave acetate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- 15 mg Anecortave Acetate (Experimental): Anecortave Acetate Sterile Suspension, 30 mg/mL, one injection of 0.5 mL in the study eye every 6 months for 48 months
  Interventions: Drug: Anecortave Acetate Sterile Suspension, 30 mg/mL
- 30 mg Anecortave Acetate (Experimental): Anecortave Acetate Sterile Suspension, 60 mg/mL, one injection of 0.5 mL in the study eye every 6 months for 48 months
  Interventions: Drug: Anecortave Acetate Sterile Suspension, 60 mg/ML
- Anecortave Acetate Vehicle (Sham Comparator): Anecortave Acetate Vehicle, one sham injection in the study eye every 6 months for 48 months
  Interventions: Other: Anecortave Acetate Vehicle

INTERVENTIONS:
Drug: Anecortave Acetate Sterile Suspension, 30 mg/mL — Posterior juxtascleral administration of suspension
  Arms: 15 mg Anecortave Acetate
Drug: Anecortave Acetate Sterile Suspension, 60 mg/ML — Posterior juxtascleral administration of suspension
  Arms: 30 mg Anecortave Acetate
Other: Anecortave Acetate Vehicle — Sham posterior juxtascleral administration of suspension
  Arms: Anecortave Acetate Vehicle

SUMMARY:
The purpose of this study was to demonstrate that Anecortave Acetate for Depot Suspension (15 mg or 30 mg) is safe and effective in arresting the progression of non-exudative (dry) age-related macular degeneration in patients who are at risk for progressing to exudative (wet) age-related macular degeneration.

ELIGIBILITY:
Inclusion Criteria:

* Dry AMD in study eye, Wet AMD in non-study eye;
* Other protocol-defined inclusion criteria may apply.

Exclusion Criteria:

* Under 50;
* Other protocol-defined exclusion criteria may apply.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2005-05; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with sight-threatening CNV in study eye | Month 48

SECONDARY OUTCOMES:
Time to development of sight-threatening CNV | Up to 48 months
Proportion of patients with stable vision | Up to 48 months

CONTACTS AND LOCATIONS:
Overall Officials: Terry Wiernas, PhD, Study Director — Study Director
Locations (1):
- Contact Alcon Call Center for Trial Locations, Fort Worth, Texas, United States